CLINICAL TRIAL: NCT00257088
Title: Prevention Services in Schools for Early Drug Abuse Risk
Brief Title: The Whole Day First Grade Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Institutes for Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA015409 (NIH); R01DA019984-01 (NIH)
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2005-08

CONDITIONS: Prevention of Drug Abuse and Dependency; Alcohol Abuse and Dependency; High Risk Sex Behavior; Smoking Tobacco; School Failure
Keywords: development; epidemiology; risk factors; randomized field trials
MeSH Terms: conditions — Alcoholism; Smoking

INTERVENTIONS:
Behavioral: whole day first grade program

SUMMARY:
This five-year prevention services application is concerned with preventing substance abuse, comorbid mental and behavioral disorders, and school failure. We will direct an integrated set of first grade classroom based preventive interventions at two correlated and confirmed early antecedents: early aggressive, disruptive behavior and poor achievement. We will test a comprehensive Whole Day (WD) program directed at improving: 1) teacher's classroom behavior management; 2) family/classroom partnerships regarding homework and discipline; and 3) teacher's instructional practices regarding academic subjects, particularly reading. We will test WD effectiveness in a developmental epidemiological design in which children and teachers are randomly assigned to intervention and standard setting (control) classrooms in 2 classrooms in each of 12 schools. While following the first grade children to the end of third grade, we will follow their first grade teachers over two subsequent cohorts of first graders to test whether the support and training structure sustains high levels of WD practice. We will also test whether the support and training structure is successful in training non-WD teachers. This prevention services aim will be augmented by an economic analysis of the costs and cost-effectiveness of the WD program. This combined services and prevention research should increase the efficiency of developing evidence-based programs and extending their use system-wide in both the prevention and education fields. The aims of our proposed work are to: 1) Implement and evaluate the effectiveness of a whole-day preventive intervention program for first-grade (WD) directed at known antecedent risk factors for later substance abuse, school failure, and comorbid mental and behavioral disorders; 2) Measure the variation in impact of WD due to variation in the experimentally manipulated quality of teachers' specific WD practices around classroom behavior management, family/classroom partnership, and quality of instruction, regarding reading, taking into account family, peer, and community factors; 3) Test effective- ness of the support structure required to sustain, and extend to other teachers high quality implementa- tion of WD; 4) Carry out economic analyses of the costs of implementing WD and their cost-effectiveness.

DETAILED DESCRIPTION:
This five-year application is concerned with preventing substance abuse, comorbid mental and behavioral disorders, and school failure. We will direct an integrated set of previously tested preventive first-grade interventions at two correlated and confirmed early antecedents: early aggressive, disruptive behavior and poor achievement. The interventions we propose to integrate and test are directed at improving: 1) teacher's classroom behavior management; 2) family/classroom partnerships regarding homework and discipline; and 3) teacher's instructional practices regarding academic subjects, particularly reading. The combined preventive and educational intervention strategy will be a single Whole Day (WD) first-grade classroom program, built on the empirically determined recognition of the interdependence of these risk factors across substance abuse and educational failure. As in our past Baltimore preventive trials, we propose to test the effectiveness of WD in a developmental epidemiological design in which children and teachers are randomly assigned to intervention and standard setting conditions (controls; SC). A special aspect of this proposal is that in the same design we propose laying a foundation for moving what we have learned into policy and practice. While following the first-grade children as far as the end of third grade, we will follow their first grade teachers over two subsequent cohorts of first graders, to test whether the support and training structure sustains high levels of WD practice. We will also test whether the support and training structure is successful in training non-WD teachers, as far as the trial results warrant. This prevention services aim will be augmented by an economic analysis of the costs and effectiveness of the WD program. The research on effectiveness combined with research on moving from effectiveness to practice should increase the efficiency of developing evidence-based programs faster and earlier in both the prevention and education fields.

This grant would set the foundation for grants for following the cohort of study children and teachers periodically to assess the preventive impact of the interventions on later substance abuse and on extending teachers' use of WD practices. This prevention research in Baltimore continues under the aegis of our Community and Institutional Board (see letters of support). This proposal involves a close institutional collaboration among the American Institutes for Research (AIR); Baltimore City Public School System (BCPSS); Morgan State University (MSU); the Oregon Social Learning Center (OSLC); the Prevention Science and Methodology Group (PSMG); the Johns Hopkins Bloomberg School of Public Health; and the Center for Academic and Reading Skills at the University of Texas-Houston.

The aims of our proposed work are to

1. Implement and evaluate the effectiveness of a whole-day preventive intervention program for first grade (WD) directed at reducing the antecedent risk factors for later substance abuse, comorbid mental and behavioral disorders, and school failure.
2. Measure the variation in the impact of WD owing to variation in the experimentally manipulated quality of teachers' specific WD practices around classroom behavior management, family/classroom partnership, and quality of instruction, particularly regarding reading. These analyses will include other sources of variation as well, in the child and in the social contexts of family, classroom and school, peers, and community.
3. Test the effectiveness of the support and training structure required to develop and maintain high-quality implementation of WD a) during the effectiveness trial; then b) as the results warrant, sustaining high-quality WD in consecutive cohorts of first graders; and then c) extending the hypothesized higher quality of WD to other than WD teachers.
4. Carry out economic analyses of the costs of implementing WD and their cost-effectiveness compared with SC with respect to reductions in risk factors for illicit substance abuse, as well as tobacco, HIV, school failure, and comorbid mental and behavioral disorders.

B. Background and Significance Over the past three decades, evidence from developmental epidemiological studies has consistently identified specific antecedent risk factors at least as early as first grade as predictive of later substance abuse and comorbid mental and behavioral disorders during the middle school years and beyond (Cairns, Cairns, & Neckerman, 1995; Farrington, 1995; Hawkins, Catalano, & Miller, 1992; Hawkins, Doueck, & Lishner, 1988; Kellam, Brown, Rubin, & Ensminger, 1983; Reid, 1993; Reid & Eddy, 1997). Many of these antecedents are exhibited in the school setting, such as aggressive, disruptive behavior in first grade and its strong correlate, poor academic achievement. These early risk factors can lead to later substance abuse and school dropout, which have considerable economic, social, and psychological consequences (Dishion, Capaldi, & Yoerger, 1999; Eddy, Reid, & Fetrow, 2000; Hawkins et al., 1992; Kellam et al., 1983; Kellam, Mayer, Rebok, & Hawkins, 1998; Maguin & Loeber, 1996; Mrazek & Haggerty, 1994; Reid, Eddy, Fetrow, & Stoolmiller, 1999 [see Appendix-1 for paper]). These risk factors are also strongly related to a host of other risk factors that separately or together are predictive during adolescence and young adulthood of not only drug abuse, but also conduct disorders and violence, depression, school drop out, and high-risk sexual behaviors. Ineffective parenting around discipline and homework; classrooms with high levels of aggressive, disruptive behavior; antisocial classmates and peers; poverty at the family level and at the school and community levels, and individual differences such as sensation seeking (Wills, Sandy, & Yaeger, 2000; Palmgreen, Donohew, Lorch, Hoyle, & Stephenson, 2001)-all have been found to increase the risk of drug abuse and related comorbid problems (Ary et al., 1999; Dishion et al., 1999; Kellam, Ling, Meriska, Brown, & Ialongo, 1998 [see Appendix-2 for paper]; Reid, Patterson, & Snyder, in press).

In Baltimore, in Oregon, and elsewhere, rigorous, developmental, epidemiologically based, randomized field trials have directed interventions at decreasing the early risk factors in the classroom, family, and peer-group settings. These trials indicate that school-based universal interventions (i.e., those addressing all children, not merely those at higher risk) can have short-term beneficial effects on aggressive behavior and achievement (Dolan et al., 1993; Ialongo et al., 1999; Reid, et al., 1999), off-task behavior (Brown, 1994a, 1993b), and depressive symptoms (Kellam, Rebok, Mayer, Ialongo, & Kalodner, 1994). Impact from first grade interventions to reduced aggression in middle school has been reported (Kellam, Rebok, Ialongo, & Mayer [see Appendix-3 for paper], 1994; Kellam, Ling et al., 1998), and delinquency (Eddy et al., 2000). Longer-term effects on illicit drug use have been observed in the Baltimore work (see Figure 1). Reductions in the initiation of tobacco use have been shown as a result of the Baltimore first grade preventive interventions in three separate cohorts (Kellam & Anthony, 1998 [see Appendix-4 for paper]; Storr, Ialongo, Kellam, & Anthony, in press). Longer-term impact has been reported in meta-analyses on illicit drug use by Nan Tobler and colleagues (1986; 2000; Tobler et al., 2000) plus other meta-analyses (Derzon & Lipsey, 1999; Gorman, 1995). Higher-fidelity implementation of the interventions also led to higher impact (Ialongo et al., 1999 [see Appendix-5 for paper], Ialongo, Poduska, Werthamer, & Kellam, 2001 [see Appendix-6 for paper]). Further, we have found compelling evidence that these universal interventions often have the greatest impact on those at highest risk of substance abuse and aggression (Brown & Liao, 1999 [see Appendix-7 for paper]; Curran & Muthèn, 1999; Muthèn & Curran, 1997; Muthèn et al., submitted; Stoolmiller, Eddy, & Reid, 2000 [see Appendix-8 for paper]).

ELIGIBILITY:
Inclusion Criteria:

Must be a first grade child in regular first grade classrooms in 12 schools in 2 academic areas of Baltimore City Public School System

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 2003-09

PRIMARY OUTCOMES:
independent observation of behavior and psychological Dx test performance
ratings by teachers and others
school records
juvenile justice records

CONTACTS AND LOCATIONS:
Overall Officials: Sheppard G Kellam, M.D., Principal Investigator — American Institutes for Research; Jeanne M Poduska, ScD, Study Director — American Institutes for Research; C. Hendricks Brown, PhD, Study Chair — University of South Florida; John B. Reid, PhD, Study Chair — Oregon Social Learning Center
Locations (1):
- AIR Center for Integrating Education and Prevention Research in Schools, Baltimore, Maryland, United States

REFERENCES:
- [Background] Storr CL, Ialongo NS, Kellam SG, Anthony JC. A randomized controlled trial of two primary school intervention strategies to prevent early onset tobacco smoking. Drug Alcohol Depend. 2002 Mar 1;66(1):51-60. doi: 10.1016/s0376-8716(01)00184-3. PMID 11850136
- [Background] Ialongo N, Poduska J, Werthamer L, and Kellam S. The Distal Impact of Two First-Grade Preventive Interventions on Conduct Problems and Disorder in Early Adolescence. Journal of Emotional & Behavioral Disorders 9(3), 146. 2001.
- [Background] Ialongo NS, Werthamer L, Kellam SG, Brown CH, Wang S, Lin Y. Proximal impact of two first-grade preventive interventions on the early risk behaviors for later substance abuse, depression, and antisocial behavior. Am J Community Psychol. 1999 Oct;27(5):599-641. doi: 10.1023/A:1022137920532. PMID 10676542
- [Background] Crijnen, Alfons A. M., Feehan, Michael, and Kellam, Sheppard G. The course and malleability of reading achievement in elementary school: The application of growth curve modeling in the evaluation of a mastery learning intervention. Learning & Individual Differences 10(2), 137. 1998. Elsevier Science Publishing Company, Inc.
- [Background] Kellam SG, Anthony JC. Targeting early antecedents to prevent tobacco smoking: findings from an epidemiologically based randomized field trial. Am J Public Health. 1998 Oct;88(10):1490-5. doi: 10.2105/ajph.88.10.1490. PMID 9772850
- [Background] Kellam SG, Ling X, Merisca R, Brown CH, Ialongo N. The effect of the level of aggression in the first grade classroom on the course and malleability of aggressive behavior into middle school. Dev Psychopathol. 1998 Spring;10(2):165-85. doi: 10.1017/s0954579498001564. PMID 9635220
- [Background] Rebok GW, Hawkins WE, Krener P, Mayer LS, Kellam SG. Effect of concentration problems on the malleability of children's aggressive and shy behaviors. J Am Acad Child Adolesc Psychiatry. 1996 Feb;35(2):193-203. doi: 10.1097/00004583-199602000-00013. PMID 8720629
- [Background] Kellam SG, Rebok GW, Ialongo N, Mayer LS. The course and malleability of aggressive behavior from early first grade into middle school: results of a developmental epidemiologically-based preventive trial. J Child Psychol Psychiatry. 1994 Feb;35(2):259-81. doi: 10.1111/j.1469-7610.1994.tb01161.x. PMID 8188798
- [Background] Kellam SG, Rebok GW, Mayer LS, Ialongo N: Depressive symptoms over first grade and their response to a developmental epidemiologically based preventive trial aimed at improving achievement. Development & Psychopathology 1994; 6:463-481
- [Background] Dolan LJ, Kellam SG, Brown CH, Werthamer-Larsson L: The short-term impact of two classroom-based preventive interventions on aggressive and shy behaviors and poor achievement. Journal of Applied Developmental Psychology 1993; 14:317-345
- [Background] Kellam SG, Anthony JC, Brown CH, Dolan L, Werthamer-Larsson L, Wilson R. Prevention research on early risk behaviors in cross-cultural studies in Needs and prospects of child and adolescent psychiatry Edited by Schmidt MH, Remschmidt H. Hogrefe & Huber Publishers, 1989
- [Background] Kellam SG, Langevin DJ. A framework for understanding "evidence" in prevention research and programs. Prev Sci. 2003 Sep;4(3):137-53. doi: 10.1023/a:1024693321963. PMID 12940466
- [Derived] Wilcox HC, Petras H, Brown HC, Kellam SG. Testing the Impact of the Whole-Day Good Behavior Game on Aggressive Behavior: Results of a Classroom-Based Randomized Effectiveness Trial. Prev Sci. 2022 Aug;23(6):907-921. doi: 10.1007/s11121-022-01334-y. Epub 2022 Mar 1. PMID 35230615
- [Derived] Poduska J, Kellam S, Brown CH, Ford C, Windham A, Keegan N, Wang W. Study protocol for a group randomized controlled trial of a classroom-based intervention aimed at preventing early risk factors for drug abuse: integrating effectiveness and implementation research. Implement Sci. 2009 Sep 2;4:56. doi: 10.1186/1748-5908-4-56. PMID 19725979